CLINICAL TRIAL: NCT04496960
Title: Safety of Tofacitinib, an Oral Janus Kinase Inhibitor, in Primary Sjogren's Syndrome; a Phase Ib-IIa Placebo-controlled Clinical Trial and Associated Mechanistic Studies
Brief Title: Safety of Tofacitinib, an Oral Janus Kinase Inhibitor, in Primary Sjogren's Syndrome
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200131; 20-D-0131
Record Dates: First submitted 2020-08-02; First posted 2020-08-04 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12-03

CONDITIONS: Sjogren's Syndrome
Keywords: Salivary; Dry Mouth; Safety; Inflammation; Xerostomia
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia; Inflammation | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: Tofacitinib (Experimental): Sjogren's Disease (SjD) patients with mild to moderate disease activity receive tofacitinib 5 mg orally twice daily for 168 days.
  Interventions: Drug: tofacitinib
- Placebo (Placebo Comparator): Sjogren's Disease (SjD) patients with mild to moderate disease activity receive placebo orally twice daily for 168 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: tofacitinib — XELJANZ(R) is the citrate salt of tofacitinib. Tofacitinib citrate is a white to off-white powder. XELJANZ(R) is supplied for oral administration as 5 mg tofacitinib (equivalent to 8 mg tofacitinib citrate) white round, immediate-release film-coated tablet.
  Other Names: Xeljanz
  Arms: Drug: Tofacitinib
Other: Placebo — white, round, film-coated tablet
  Arms: Placebo

SUMMARY:
Background:

An autoimmune disease is one in which the immune system attacks a person's own body. Sjogren's syndrome (SS) is an autoimmune disease. It often involves multiple systems and organs of the body. Researchers are trying to find new, more effective and safe treatments for SS.

Objective:

To evaluate the safety and tolerance of tofacitinib in people with SS.

Eligibility:

Adults ages 18-75 with SS.

Design:

Participants will be screened on a separate protocol. They will undergo:

* Medical and dental history
* Physical exam
* Medicine review
* Electrocardiogram to test the heart s electrical activity (Participants will lay on a table. Sticky pads will be placed on their body.)
* Eye exam and test for dry eyes
* Oral, head, and neck exams
* Plaque collection (Dental plaques and tongue and mucosal scrapings will be collected using a small tongue depressor.)
* Salivary gland ultrasound
* Blood and urine tests
* Minor salivary gland biopsy (The lower lip will be numbed. Several tiny salivary glands will be removed through a small incision.)
* Saliva collection
* Disease assessment.

Participants will repeat some of the screening tests during the study.

Participants will take capsules of the study drug or a placebo by mouth for 168 days.

Participants will have tests to measure blood pressure and the speed of blood flow through the organs. They will also have a test that examines the function and reaction of the blood vessels. For these tests, they will wear blood pressure cuffs and other sensors.

Participants will complete questionnaires about their health.

Participants will have 9 study visits over 28 weeks. They may be contacted by phone between study visits.

DETAILED DESCRIPTION:
Study Description:

As a primary objective, this study represents an innovative investigative measure of the safety and tolerability of JAK inhibition in participants with primary Sjogren's syndrome. Secondary objectives will include investigating the effects of Tofacitinib on target tissues (e.g., salivary glands), systemic inflammation, and on vascular function in SS participants. We also aim to identify biomarkers of response that may be useful as endpoints in future studies.

Objectives:

Primary Objective:

-To determine the safety and tolerability of Tofacitinib in participants with SS and mild to moderate disease activity.

Secondary Objectives:

* To assess clinical improvement after treatment with Tofacitinib as measured by changes in the European League Against Rheumatism (EULAR) Sjogren's syndrome Disease Activity Index (ESSDAI) and no worsening on the Physician s Global assessment Scale (PGA).
* To demonstrate that treatment with Tofacitinib is effective clinically and biologically in SS individuals with mild to moderate disease.
* To investigate the effects of Tofacitinib on systemic biomarkers of SS as measures biological effects that can be used as outcome measures to power a larger Clinical Trial.

Endpoints:

Primary Endpoint:

-Safety and tolerability will be measured by assessment of adverse events (AEs) and clinical safety laboratory tests throughout the study. Toxicity is defined as any study drug-related Grade 3 adverse event or higher (as measured by the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0).

Secondary Endpoints:

Preliminary assessments of clinical response will be measured by:

* Changes in the ESSDAI score between Baseline and Day 168 (end of treatment)
* Changes in the Physician's Global Assessment (PGA) scores between baseline and study day 168.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult primary SS participants with mild-to-moderate disease activity will be eligible for this study. Enrolled participants can be naïve or failed immunosuppressive therapy beyond antimalarials and glucocorticoids; to prevent bias in the cohort of participants with more recalcitrant disease. We expect that Tofacitinib is a potential second line therapy, in addition to antimalarials and glucocorticoids, depending on the participant's initial presentation and response. Women and members of minority groups, if eligible, will be included in accordance with the NIH Policy on Inclusion of Women and Minorities as Participants in Research Involving Human Participants.

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability of participant to understand and the willingness to sign a written informed consent document.
2. Participation and enrollment in companion protocol, 15-D-0051, Characterization of Diseases with Salivary Gland Involvement.
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Male or female, aged between 18-75 years
5. In good general health as evidenced by medical history
6. Meets the 2002 American European Consensus Group classification criteria for primary Sjogren's Syndrome or 2016 American College of Rheumatology/European League against Rheumatism Classification Criteria (ACR-EULAR) with mild to moderate disease activity defined as ESSDAI between 0 to 13 at the screening visit and >0 ml/min/gland stimulated saliva flow.
7. Ability to take oral medication and be willing to adhere to the study intervention regimen
8. If on glucocorticoids, the dose must be less than 10 mg daily and stable for the 4 weeks (28 days) prior to screening visit.
9. If on hydroxychloroquine or other antimalarials such as chloroquine or quinacrine, the dose must have been stable for the 12 weeks (96 days) prior to screening visit. The maximum allowed dose is hydroxychloroquine up to 400 mg/day or 6.5 mg/kg/day if more than 400 mg/day. The maximum allowed dose for chloroquine phosphate is up to 500 mg daily and for quinacrine up to 100 mg daily.
10. Participants may be on lipid lowering medications if initiated at least 3 months prior to the screening visit and dose must be stable for 4 weeks (28 days) prior to study entry.
11. Males and females with potential for reproduction must agree to practice effective birth control measures. Females should be on adequate contraception if they are of child-bearing potential documented by a clinician, unless participants or spouse have previously undergone a sterilization procedure. Adequate birth control measures are: intrauterine device (IUD) alone or hormone implants, hormone patches, injectable, or oral contraceptives plus a barrier method (male condom, female condom or diaphragm), abstinence or a vasectomized partner.
12. Agreement to adhere to Lifestyle Considerations throughout study duration

EXCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must not meet any of the following criteria:

1. Current or prior treatment with rituximab, belimumab or any other biologic agent in the 6 months prior to screening.
2. Current treatment with methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus, or other less common immunomodulatory drugs such as those falling into the class of disease-modifying antirheumatic drugs (DMARDs), not otherwise specified herein. Participants previously on methotrexate, azathioprine, mycophenolate mofetil, cyclosporine or tacrolimus, or other DMARDs should have withdrawn drug for at least 8 weeks (56 days) at the time of screening.
3. Treatment with cyclophosphamide, pulse methylprednisolone or IVIG within 6 months prior to screening.
4. Current treatment with potent inhibitors of Cytochrome P450 3A4 (CYP3A4) (e.g., ketoconazole) or receiving one or more concomitant medications that result in both moderate inhibition of CYP3A4 and potent inhibition of CYP2C19 (e.g., fluconazole) that would increase serum availability of Tofacitinib. Past treatment with the aforementioned agent is allowed if it was more than a week prior to the administration of the first dose of study medication.
5. History of chronic liver disease, not including well-controlled Sjogren's-related chronic liver disease or elevated liver function tests (LFT):

   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >= 2x upper limit of normal at screening
   * Serum unconjugated bilirubin > 2mg/dL at screening
6. Serum creatinine >1.5mg/dL.
7. Protein to creatinine ratio of more than 1mg/dL at screening (repeated and confirmed three times or confirmed with 24 hours urine protein of more than 1000mg).
8. Active urinary sediment (WBC, red blood cell (RBC) or mixed cellular casts 1+ or more /hpf)).
9. Hypercholesterolemia: Values after 8-12 hour fasting blood specimen: total cholesterol >250 mg/dL or LDL >180 mg/dL or hypertriglyceridemia (triglyceride >300 mg/dL) within-45 days of screening visit.
10. WBC <2500/microliter or absolute neutrophil count (ANC) <1,000/microliter, Hgb <9.0 g/dL or platelets <70,000/microliter or absolute lymphocyte count < 500/microliter.
11. Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test at screening.
12. A history of drug or alcohol abuse within the 6 months prior to screening.
13. Currently receiving hemodialysis, peritoneal dialysis, or intestinal dialysis.
14. Active infection that requires the use of oral or intravenous antibiotics unresolved at least 14 days prior to the administration of the first dose of study medication.
15. Active chronic infections including but not limited to HIV, Hepatitis B, Hepatitis C, and BK viremia at screening visit.
16. Current or previous diagnosis of malignant disease, except for basal cell or squamous cell carcinoma of the skin with complete excision and clear borders or adequately treated in situ carcinoma of the cervix.
17. Known active tuberculosis. Participants with treated latent tuberculosis (LTB) will be eligible to participate. Participants with untreated LTB will not be excluded but will be evaluated by an infectious disease (I.D.) consultant and may become eligible for trial based on infectious disease consultant recommendations.
18. History of severe or systemic infection caused by common pathogens, or history of infection with pathogens that normally do not cause human disease.
19. Participants with active renal or central nervous system disease or a high activity level in any organ system (except articular) in ESSDAI.
20. Participants with known increased risk factors for major adverse cardiac event (MACE) including a history of:

    * Ischemic heart disease (e.g., history of acute myocardial infarction)
    * Heart failure
    * Cardiomyopathy
    * Severe valvular heart disease
    * Significant arrhythmias
    * Chronic renal failure
    * Cerebrovascular accident or transient ischemic attack
    * Uncontrolled diabetes mellitus
    * Uncontrolled hypertension
    * Current smokers or former smokers with less than 3 years since complete cessation and/or >20 pack-years of smoking history.
21. Significant impairment of major organ function (lung, heart, liver, kidney) or any condition that, in the opinion of the Investigator, would jeopardize the participant's safety following exposure to the study drug.
22. Known history of arterial or venous thrombosis or at high risk for clotting disorder
23. Psychiatric illness or history of medical non-compliance that the study team feels will make the patient unlikely to complete the study
24. Uncontrolled thyroid disease as per PI or medically responsible investigator.
25. Known allergic reactions to Tofacitinib or its components
26. Treatment with another investigational drug/intervention within six months except for COVID-19 vaccines or therapies that have been granted an FDA emergency authorization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2026-09-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Blake M Warner, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Study complies with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule.
Time Frame: At the time of publication or after 3 years, which ever comes first.
Access Criteria: NIH's policy for data-sharing for federally funded genome-wide association studies requires that genotypic and phenotypic information from such studies will be made available through the NIH data repository. Only coded de-identified data will be available.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-D-0131.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 Participants were consented
  * 12 participants started the study
  * 11 participants were screen failure
Period: Overall Study
Arm/Group | Drug: Tofacitinib | Placebo
Started | 8 | 4
Completed | 8 | 3
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Tofacitinib | Placebo | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events by Grade/Category
Description: Count of adverse events by grade was assessed using the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
  Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental ADL.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4: Life-threatening consequences; urgent intervention indicated.
  Grade 5: Death related to adverse event.
  Serious is defined as any grade 3 or higher adverse event.
  Toxicity is defined as any study drug-related Grade 3 or higher adverse event.
Time Frame: Up to day 196
Population: Intent to treat population
Measure: Number; unit: Count of adverse events
Units Other Than Participants: Count of adverse events
Arm/Group | Drug: Tofacitinib | Placebo
Number analyzed (Participants) | 8 | 4
Number analyzed (Count of adverse events) | 33 | 12
Count of adverse events
  Grade 1 | 19 | 3
  Grade 2 | 10 | 7
  Grade 3 | 4 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0
  Serious | 4 | 1
  Toxicity | 4 | 0

2. Primary Outcome: Participants With Adverse Events
Description: Number participants with any adverse events by grade and severity was assessed using the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activity of daily living (ADL).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to adverse event.
  Serious is defined as any grade 3 or higher adverse event.
  Toxicity is defined as any study drug-related Grade 3 or higher adverse event.
Time Frame: Up to day 196
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Tofacitinib | Placebo
Number analyzed (Participants) | 8 | 4
Participants
  Subjects with at least one adverse event | 7 | 3
  Subjects with at least one adverse event with grade 3 and above | 1 | 1
  Subjects with at least one Severe adverse event (SAE) | 1 | 1
  Subjects with at least one toxicity | 1 | 0

3. Secondary Outcome: Change in Physicians Global Assessment (PGA) Score
Description: The Physician Global Activity (PGA) is a subjective physician reported disease activity index that uses a 10-cm Visual Analog Scale (VAS) to score a patient's disease activity. The 10-cm visual analogue scale (VAS) was scored by a physician with a vertical line on the scale marking disease activity where 0 cm indicates no evidence of disease activity, and 10 cm indicates severe disease activity, with score reported on a scale from 0-10. Higher score indicates more disease activity. Change in disease activity index was measured as the mean difference in disease activity scores between time points. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Time Frame: Day 168 minus day 1
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Drug: Tofacitinib | Placebo
Number analyzed (Participants) | 8 | 3
Units on a scale | 0 (3.07) | -1.67 (2.89)

4. Secondary Outcome: Change in EULAR Sjögren's Syndrome (SS) Disease Activity Index (ESSDAI) Score
Description: The EULAR Sjögren's syndrome (SS) disease activity index (ESSDAI) is a systemic disease activity index designed to measure disease activity in patients with primary SS. It includes 12 organ domains (e.g., constitutional, glandular, neurological) for disease activity, each with a 4-point scale (0 = No activity; 3=High activity). These scores are then multiplied by domain-specific weights (1-6) and summed to produce a total score ranging from 0 to 123, with higher scores indicating greater disease activity. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Time Frame: Day 168 minus day 1
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Drug: Tofacitinib | Placebo
Number analyzed (Participants) | 8 | 3
Units on a scale | -0.13 (1.13) | -1.33 (2.31)

5. Secondary Outcome: Change in Whole Unstimulated Saliva Flow
Description: Changes in salivary flow was assessed by measuring whole unstimulated saliva flow (WUS) and glandular parotid and submandibular/sublingual unstimulated and 0.2% citric acid stimulated flow rates using ultrasonograph. Validated scoring criteria was used to assess ultrasonographic feature parameters at baseline and at the study day 168. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Time Frame: Day 168 minus day 1
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: ml/min/gland
Arm/Group | Drug: Tofacitinib | Placebo
Number analyzed (Participants) | 8 | 3
ml/min/gland | -0.13 (1.13) | -1.33 (2.31)

6. Secondary Outcome: Change in Whole Stimulated Saliva Flow
Description: Changes in salivary flow was assessed by measuring whole stimulated saliva flow and glandular parotid and submandibular/sublingual stimulated and 0.2% citric acid stimulated flow rates using ultrasonograph. Validated scoring criteria was used to assess ultrasonographic feature parameters at baseline and at the study day 168. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Time Frame: Day 168 minus day 1
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: ml/min/gland
Arm/Group | Drug: Tofacitinib | Placebo
Number analyzed (Participants) | 8 | 3
ml/min/gland | 10.6 (1.13) | 6.21 (2.31)

7. Secondary Outcome: Change in EULAR Sjögren's Syndrome (SS) Patient Reported Index (ESSPRI)
Description: The EULAR Sjögren's Syndrome (SS) Patient Reported Index (ESSPRI) is a patient-reported outcome measure (PROM) that focuses on the subjective experience of symptoms in SS. The tool assesses the key symptoms of dryness, pain and fatigue. A single 0-10 numerical scale is used to assess each of these symptoms. Final score is the average of the scores from the three domains. A final ESSPRI score of less than 5 is considered indicative of acceptable disease status, while a score of 5 or higher suggests high disease activity. Questionnaire was completed at baseline and day 168. Data was analyzed as
Time Frame: Day 168 minus day 1
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Drug: Tofacitinib | Placebo
Number analyzed (Participants) | 8 | 3
Units on a scale | -1.33 (2.04) | 0.78 (0.51)

ADVERSE EVENTS:
Time Frame: Up to day 196
Arm/Group | Drug: Tofacitinib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/3
Other Adverse Events (participants affected / at risk) | 6/8 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: Tofacitinib (N=8) | Placebo (N=3)
Neutrophil count decreased (Investigations) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: Tofacitinib (N=8) | Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 1
BK virus infection (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Barotrauma (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04496960/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT04496960/ICF_002.pdf